CLINICAL TRIAL: NCT03262883
Title: The Prevalence of Chronic Critical Illness Adult Intensive Care Units in Turkey
Brief Title: The Prevalence of Chronic Critical Illness in Turkey
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Collaborators: Kahramanmaras Sutcu Imam University (Other); Izmir Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hilmi Demirkiran, MD, Assistant Professor, Yuzuncu Yil University
Other Study IDs: Chronic critical illness
Record Dates: First submitted 2017-08-18; First posted 2017-08-25 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Chronic Critical Illness
Keywords: Prolonged akut mechanical ventilation; Tracheotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Critical Illness: The patients who is over 18 years old and staying in the critical care unit at least 8 days. Additional criterias:
  1. Prolonged mechanical ventilation (longer than 96 hours)
  2. Tracheostomy
  3. Sepsis
  4. Serious injury (burn)
  5. Stroke (hemorhagic or ischemic)
  6. Traumatic brain injury

SUMMARY:
It is known that the number of Chronic Critical İllnes, an iatrogenic condition, increases all over the world. The prevalence of Chronic Critical Illness in Turkey is unknown. The investigators aimed to evaluate the etiology, comorbid conditions, demographic data, prevalence, mortality and costs of these patient in intensive care units in Turkey. In this multi-centered study, The investigators will retrospectively review the last 1 year of patients receiving treatment at the Adult Intensive Care Unit.

DETAILED DESCRIPTION:
The patients who survive an acute critical illness in the Intensive Care Unit (ICU) may be delayed in a situation where they are sometimes totally independent before hand due to iatrogenic causes such as infections, dysfunctions, psychological disorders. This can take weeks, sometimes months. This disease is called "Chronic Critical Illness" (CCI).

Most researchers associate CCI with the need for prolonged acute mechanical ventilation or the opening of tracheostomy for prolonged acute mechanical ventilation. There is no single condition that does not require an extended mechanical ventilation from CCI. In conclusion, CCI is characterized by long-term care requiring survival and it is predicted that the cost of these patients will increase with the new patients whose cost will be added in the coming years. In the United States, the number of CCI is around 250,000, and this figure has increased by 50-100% in the last 10 years. At least 50% of these patients die in one year and less than 12% recover and become discharged. The annual cost of these patients' health care system is over $ 20 billion. The prevalence of CCI in Turkey is still unknown. In this study, it was aimed to investigate the prevalence of patients with Chronic Critical Syndrome in intensive care units in Turkey.

ELIGIBILITY:
Inclusion Criteria:

The patient who is over 18 years old, taking mechanical ventilation support and staying in the critical care unit at least 8 days. Additional criterias; Clinical diagnosis of following situations:

1. Prolonged mechanical ventilation
2. Tracheotomia
3. Sepsis
4. Serious injury (burn)
5. Stroke ( hemorhagic or ischemic)
6. Traumatic brain injury

Exclusion Criteria:

1. The patients who not having mechanical ventilation support
2. The patient staying less than 8 days in the intensive care unit
3. The patient younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient older than 18 years old staying in the intensive care unit longer than 8 days
Sampling Method: Probability Sample
Enrollment: 2493 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-04-28 (Actual)

PRIMARY OUTCOMES:
Critical care unit mortality | 30 day and 90 day
  The mortality change rates in the 30th days and 90th days

SECONDARY OUTCOMES:
Critical care unit costs | Duration of intensive care unit stay (8 day after the hospitalisation to sixth month)
  Costs of patients staying in the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Hilmi Demirkıran, Principal Investigator — Official of the university
Locations (1):
- Yuzuncu Yıl University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided